CLINICAL TRIAL: NCT04357574
Title: Assessing the Provider Implementation and Experience of TeleHealth During COVID-19 and Impact on Acute Encounters
Brief Title: Assessing the System for High-Intensity Evaluation During Radiotherapy During Changes in Response to COVID-19
Acronym: CORONA-SHIELD
Status: Enrolling by invitation | Type: Observational
Sponsor: Duke University (Other)
Collaborators: University of California, San Diego (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00105266
Record Dates: First submitted 2020-04-20; First posted 2020-04-22 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: COVID-19; Cancer
MeSH Terms: conditions — COVID-19; Neoplasms | interventions — Telemedicine

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Radiation Oncology Providers: Faculty physicians, residents and advanced practice providers in the Radiation Oncology Department in Duke University Health System (DUHS)
  Interventions: Other: Telehealth

INTERVENTIONS:
Other: Telehealth — patients have virtual visits with Radiation Oncology providers in lieu of in person clinic visits as a necessary response to COVID-19

SUMMARY:
The primary objective of this research study is to assess Radiation Oncology healthcare providers (i.e. faculty, residents and advanced practice providers (APPs) implementation and perception of telehealth for on treatment patients in lieu of in person on treatment visits during standard of care radiotherapy during COVID-19.

DETAILED DESCRIPTION:
A secondary aim will be to evaluate the rates of acute care during COVID-19 with telehealth in comparison to the rates during our prior Quality Improvement (QI) project (NCT04277650), considering the risk prediction based on our previously developed ML algorithm. Patient risk during this period will be assessed by the ML algorithm and actual rates of Emergency Department visits and hospitalizations (acute encounters) will be compared to the results of our prior QI project. These data will be used to discern how actual rates of acute care compare to providers' expectations both with and without telehealth implementation. Reasons for acute encounters and associated healthcare costs compared to patients undergoing standard of care assessments in NCT04277650 will be assessed to determine the percentage that are COVID-19 related. Basic demographic, disease, location of acute care, form of clinical assessments (video, in-person, telephone, etc.), and treatment information regarding the patients will also be captured following the completion of the research project for assessment.

These endpoints will establish how our current COVID-19-based precautions impact treatment-related outcomes in patient care.

ELIGIBILITY:
Inclusion Criteria:

• started outpatient radiation therapy with or without concurrent systemic therapy at Duke Cancer Center during the COVID-19 outbreak

Exclusion Criteria:

* undergoing total body radiation therapy for hematopoetic stem cell transplantation
* undergoing therapy as inpatient
* completed radiation therapy prior to algorithm execution

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing radiation therapy in the Department of Radiation Oncology at Duke Cancer Center during the COVID-19 outbreak
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2020-04-14 (Actual); Primary Completion 2027-04 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Radiation Oncology providers perception of of telehealth for on treatment patients in lieu of in person on treatment visits during COVID-19 | 12 months
  survey assessment scored as strongly agree (positive perception) through strongly disagree (negative perception)

SECONDARY OUTCOMES:
Number of missed telehealth clinical evaluation visits during COVID-19 | 12 months
Number of unplanned emergency department visits or hospital admissions during COVID-19 | 12 months
Number of acute care visits with listed reason as anemia, nutrition (including dehydration), diarrhea, emesis, infectious (including fever, pneumonia, and sepsis), nausea, neutropenia, pain category during COVID-19 | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Manisha Palta, MD, Principal Investigator — Duke Health
Locations (1):
- Duke Cancer Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No